CLINICAL TRIAL: NCT05564767
Title: Effect of Two Probiotic Formulations on Mental Health and Mood Biomarkers in Adults With Depressive Symptoms: A Pilot Randomized Placebo-controlled Trial
Brief Title: Effect of Two Probiotic Formulations on Mental Health and Mood Biomarkers in Adults With Depressive Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chr Hansen (Industry)
Responsible Party: Sponsor
Organization: ChrHansen (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HND-MH-051
Record Dates: First submitted 2022-09-29; First posted 2022-10-04 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Depression, Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- B. adolescentis Bif-038 (Experimental): Probiotic capsule (single strain)
  Interventions: Dietary Supplement: B. adolescentis Bif-038
- Lacticaseibacillus rhamnosus, LGG® and Bifidobacterium, BB-12® (Experimental): Probiotic capsule (combination strain)
  Interventions: Dietary Supplement: Lacticaseibacillus rhamnosus, LGG® and Bifidobacterium, BB-12®
- Placebo (Placebo Comparator): Placebo capsule
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: B. adolescentis Bif-038 — B. adolescentis Bif-038 (probiotic capsule) delivered orally once daily at a minimum of 5 billion CFU/day
  Arms: B. adolescentis Bif-038
Dietary Supplement: Lacticaseibacillus rhamnosus, LGG® and Bifidobacterium, BB-12® — Lacticaseibacillus rhamnosus, LGG® and Bifidobacterium, BB-12® (probiotic capsule) delivered orally once daily at a minimum of 1 billion CFU/day
  Arms: Lacticaseibacillus rhamnosus, LGG® and Bifidobacterium, BB-12®
Dietary Supplement: Placebo — Placebo capsule delivered orally once daily
  Arms: Placebo

SUMMARY:
This is a 3-arm, parallel-group, randomized, double-blind, placebo-controlled pilot trial. Sixty adults presenting with depressive symptoms will be randomly allocated to one of 3 groups comprising (1) Bifidobacterium adolescentis or (2) Lactocaseibacillus rhamnosus LGG and Bifidobacterium BB-12 or (3) a placebo for 12 weeks.

At baseline (Visit 2), midpoint (Visit 3) and end-of-study (Visit 4) visits, participants meeting eligibility criteria will complete the BDI-II, BAI, DASS-21 and PROMIS Sleep questionnaires and blood samples will be collected for biomarker assessments. Fecal samples will be collected prior to the baseline and end-of-study visits for microbial profiling.

DETAILED DESCRIPTION:
This is a 3-arm, parallel-group, randomized, double-blind, placebo-controlled pilot trial. Sixty adults presenting with depressive symptoms will be randomly allocated to one of 3 groups comprising (1) Bifidobacterium adolescentis or (2) Lactocaseibacillus rhamnosus LGG and Bifidobacterium BB-12 or (3) a placebo for 12 weeks.

At screening (Visit 1), the study design will be explained to participants, following which signed GDPR and study informed consent will be obtained. Participants will be assessed for eligibility, medical history and concomitant therapies.

At baseline (Visit 2), midpoint (Visit 3) and end-of-study (Visit 4) visits, participants meeting eligibility criteria will complete the BDI-II, BAI, DASS-21 and PROMIS Sleep questionnaires and blood samples will be collected for biomarker assessments. Fecal samples will be collected prior to the baseline and end-of-study visits for microbial profiling.

ELIGIBILITY:
Inclusion Criteria:

1. Generally healthy adults (male and female) 18 to 65 years
2. Currently experiencing depressive symptoms as indicated by a score of between 20 and 40 on the BDI-II at both the screening and baseline visit
3. Body mass index (BMI) between 18.5 and 30.0 kg/m2
4. Non-smoker
5. No plan to change dietary or exercise habits during the study period
6. No recent history (within 3 months) or plan to commence new treatments over the study period
7. Willing and able to take probiotic/placebo regimen for 12 weeks
8. Understand, willing and able to comply with all study procedures
9. Willing to provide a personally signed and dated informed consent form detailing all pertinent aspects of the trial.

Exclusion Criteria:

1. Suffering from recently diagnosed or unmanaged medical conditions including but not limited to: diabetes, hyper/hypotension, cardiovascular disease, a gastrointestinal disease requiring regular use of medications, gallbladder disease, autoimmune disease, endocrine disease, acute or chronic pain condition, or cancer/malignancy
2. Diagnosis of psychiatric or neurological conditions including but not limited to: psychiatric disorders other than mild-to-moderate depression and/or anxiety disorder, or neurological disease (e.g., Parkinson's, Alzheimer's disease, intracranial hemorrhage, head or brain injury)
3. Regular medication intake, including but not limited to anticholinergics, anti-epileptics, acetylcholinesterase inhibitors, benzodiazepines, antipsychotics, opioids, or corticosteroids.
4. Within 2 months before screening, the use of pharmaceutical medications, including but not limited to immunosuppressant drugs, antibiotics, and steroids
5. Change in medication (dose or type) in the last 3 months or an expectation to change during the study duration. Permitted medications include, but are not limited to, pharmaceutical antidepressants such as selective serotonin reuptake inhibitors (SSRIs), and serotonin and norepinephrine reuptake inhibitors (SNRIs), cholesterol-lowering medications, antihypertensives, proton pump inhibitors, and thyroid medications,
6. Use of probiotics or mood support supplement up to 4 weeks before study commencement
7. Current or 12-month history of illicit drug abuse
8. Alcohol intake greater than 14 standard drinks per week
9. Any significant surgeries over the last year
10. Women who are pregnant, breastfeeding or intend to fall pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2022-10-17 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2023-03-20 (Actual)

PRIMARY OUTCOMES:
Beck Depression Inventory-II (BDI-II) score | 12 weeks
  Change in BDI-II score after 12 weeks

SECONDARY OUTCOMES:
Beck Anxiety Inventory (BAI) score | 12 weeks
  Change in BAI score
Depression, Anxiety, Stress Scale (DASS-21) total score | 12 weeks
  Change in DASS-21 total score
DASS-21 Stress score | 12 weeks
  Change in DASS-21 Stress score
DASS-21 Depression score | 12 weeks
  Change in DASS-21 Depression score
DASS-21 Anxiety score | 12 weeks
  Change in DASS-21 Anxiety score
Brain-derived neurotrophic factor blood concentration | 12 weeks
  Change in brain-derived neurotrophic factor blood concentration

OTHER OUTCOMES:
PROMIS Sleep Disturbance and Sleep-Related Impairment Scale score | 12 weeks
  Change in PROMIS Sleep Disturbance and Sleep-Related Impairment Scale score
Tumor necrosis factor-alpha blood concentration | 12 weeks
  Change in tumor necrosis factor-alpha blood concentration
Interleukin-6 blood concentration | 12 weeks
  Change in interleukin-6 blood concentration
Interleukin-1beta blood concentration | 12 weeks
  Change in interleukin-1beta blood concentration
High sensitivity C-reactive protein blood concentration | 12 weeks
  Change in high sensitivity C-reactive protein blood concentration
Interferon-gamma blood concentration | 12 weeks
  Change in interferon-gamma blood concentration
Lipopolysaccharide-binding protein blood concentration | 12 weeks
  Change in lipopolysaccharide-binding protein blood concentration
Intestinal fatty acid-binding protein blood concentration | 12 weeks
  Change in intestinal fatty acid-binding protein blood concentration
Blood cortisol concentration | 12 weeks
  Change in blood cortisol concentration
Hair cortisol concentration | 12 weeks
  Change in hair cortisol concentration
Heart rate variability | 12 weeks
  Change in heart rate variability via electrocardiogram (ECG) measurements
Fecal microbial profile | 12 weeks
  Change in fecal microbial profile via shotgun metagenomic sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Lopresti, PhD, Principal Investigator — Clinical Research Australia
Locations (1):
- Clinical Research Australia, Duncraig, Western Australia, Australia